CLINICAL TRIAL: NCT06421402
Title: Knowledge for Improving Indoor Air Quality and Health: Follow up of 200 High-risk Chronic Respiratory Patients During 24 Months.
Brief Title: K-HEALTH in AIR - Barcelona Pilot - Cohort
Status: Enrolling by invitation | Type: Observational
Sponsor: Institut d'Investigacions Biomèdiques August Pi i Sunyer (Other)
Collaborators: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Josep Roca Torrent, Principal Investigator, Institut d'Investigacions Biomèdiques August Pi i Sunyer
Other Study IDs: HCB/2023/0126; 101057693 (Other Grant/Funding Number: HaDEA)
Record Dates: First submitted 2024-04-29; First posted 2024-05-20 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: Severe Asthma; COPD
Keywords: Prevention of Unplanned Hospital Admissions; Nurse Case Manager; COPD; Severe Asthma; Integrated Care; Digital support; Indoor Air Quality
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive | interventions — Routinely Collected Health Data

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Follow-up 200 high-risk chronic respiratory outpatients for 2 years.: The INTERVENTION (PHASE I, 2024) will have four components: i) Assessment of Lung Function Testing, ii) Monitoring of IAQ at patients' homes (and analysis of the relationships between IAQ and health events), iii) Evaluation of advanced digital support to a novel clinical process to enhance early identification and management of exacerbations (questionnaires, chat, patients' self-capturing sensors, and iv) Development, and refinement, of machine learning-based predictive modelling for supporting clinical decision making.
  During PHASE II (2025), the INTERVENTION will consist of the assessment (Quintuple Aim) of the novel integrated care service, as well as the evaluation of its potential for scalability (CFIR).
  See inclusion/exclusion criteria and planned measurements in the enclosed documents.
  Interventions: Other: Air quality monitoring at patient's home; Other: Questionnaires: Baseline & every six months; Diagnostic Test: Lung function Testing: Baseline & every six months & during exacerbations; Other: EMR & registry data; Device: Communication channel - Health Circuit Mobile App (Herranz C. JMIR 2023); Device: Physiological data - Beat One Watch; Device: Patient Empowerment; Other: Characteristics of exacerbations
- Control Group: The control group will be introduced in Phase II (2025) to estimate the potential for healthcare value generation of the novel integrated care service. It will include patients with equivalent characteristics who receive standard of care practice, without the interventions carried out in the cohort group.
  The control group will be shaped using 1-to-1 propensity score matching techniques. Data from the control group will be obtained from electronic medical records and registry information. In a randomly selected subset of 50 individuals from the control group a Quintuple Aim assessment will be done.
  Interventions: Other: EMR & registry data

INTERVENTIONS:
Other: Air quality monitoring at patient's home — Indoor Air Quality:
  - MICA-INBIOT system: temperature (ºC), humidity (%), CO2 (ppm), total Volatile Organic Ccompounds (VOCs) (ppb), Formaldehyde (µg/m3); and Particulate Matter (PM) 1/2.5/4/10 (µg/m3)
  Outdoor Air Quality:
  - Aeris Weather platform: NO, NO2, NOx, SO2, SO3, CO, and PM10, all expressed in µg/m3
  Groups: Follow-up 200 high-risk chronic respiratory outpatients for 2 years.
Other: Questionnaires: Baseline & every six months — General surveys:
  * PROMs: ICHOM Adult Set; encompassing Patient Reported Outcomes Measurement Information System (PROMIS 10), World Health Organization Wellbeing Index (WHO 5) and World Health Organization Disability Assessment Schedule (WHO-DAS 12) questionnaires.
  * PREMs: Patient-Reported Indicator Survey (PaRIS)
  Disease specific questionaires:
  * COPD: COPD Assessment Test (CAT); modified Medical Research Council (mMRC) Dyspnea scale.
  * Asthma: Asthma Control Test (ACT); Test of Adherence to Inhalers (TAI-12); Asthma Quality of Life Questionnaire (mini AQLQ); Sino-Nasal Outcome Test (SNOT-22).
  Groups: Follow-up 200 high-risk chronic respiratory outpatients for 2 years.
Diagnostic Test: Lung function Testing: Baseline & every six months & during exacerbations — * Forced Spirometry: Forced Vital Capacity (FVC) and Forced Expiratory Volume in 1 second (FEV1)
  * Forced Oscillation Technique: Impedance, resistance and reactance.
  Ancillary measurements: Systemic arterial pressure and pulse oximetry.
  Groups: Follow-up 200 high-risk chronic respiratory outpatients for 2 years.
Other: EMR & registry data — Electronic Medical Records (EMRs): Updated every twelve months to track clinical events from Hospital and Primary Care databases.
  Registry data: from the Catalan Health Surveillance System (CHSS).
Device: Communication channel - Health Circuit Mobile App (Herranz C. JMIR 2023) — Health Circuit: chat, short questionnaires (Likert scale). As needed.
  Groups: Follow-up 200 high-risk chronic respiratory outpatients for 2 years.
Device: Physiological data - Beat One Watch — Enhanced with real-time physiological data tracking (heart rate, steps walked and Heart Rate Variability (HRV))
  Groups: Follow-up 200 high-risk chronic respiratory outpatients for 2 years.
Device: Patient Empowerment — Mobile App Health Circuit: follow-up of the personalized action plan agreed with the patient & reference doctor
  Groups: Follow-up 200 high-risk chronic respiratory outpatients for 2 years.
Other: Characteristics of exacerbations — Health Circuit: home-based oscillometry, daily disease-specific questionnaire during the acute episode and continuous assessment of physiological variables.
  Groups: Follow-up 200 high-risk chronic respiratory outpatients for 2 years.

SUMMARY:
The study protocol is part of the European (EU) project "Knowledge for improving indoor AIR quality and HEALTH" (K-HEALTHinAIR, 2022-2026 - registry 101057693), which focuses on enhancing our understanding of how poor indoor air quality (IAQ) affects human health. Specifically, the project aims to identify IAQ determinants of adverse health events and to explore the development of cost-effective strategies for the precise monitoring and improvement, of IAQ across Europe.

With the current study protocol, the Barcelona Pilot, at the Integrated Health District of Barcelona-Esquerra (AISBE, 520 k citizens), is conducting a cohort study over a two-year period (January 2024 to December 2025) to explore the relationships between IAQ (assessment of chemical pollutants in patients' homes) and health status (acute episodes) in multimorbid patients with chronic respiratory diseases (asthma and Chronic Obstructive Pulmonary Disease - COPD) over a two-year period.

The protocol investigates the effectiveness of customized interventions across four critical areas: i) Advanced lung function testing, ii) Continuous IAQ monitoring, iii) Advanced digital support to innovative clinical processes, and iv) Predictive modeling for early identification and management of exacerbations. The ultimate objective is to design and evaluate an innovative integrated care service aiming at enhancing both IAQ and the management of multimorbid patients with chronic obstructive respiratory diseases, with focus on COPD and severe asthma.

DETAILED DESCRIPTION:
The study is structured as a comprehensive two-phase approach. From January to December 2024 (Phase I) the protocol focuses on the assessment, and refinement, of the four core components of the study: i) Enhanced lung function testing, ii) IAQ home monitoring, iii) Advanced digital support to innovative clinical processes, and iv) Predictive modelling for early detection and management of exacerbations. The main outcome at the end of Phase I is the design of an innovative integrated care service aiming at enhanced management of exacerbations and reduction of unplanned hospitalizations in high-risk patients.

From January to December 2025 (Phase II), the protocol aims to refine the novel clinical process, including the four core components alluded to above, as well as to evaluate the potential for healthcare value generation and scalability/transferability of the new integrated care service.

PHASE I (2024):

1. Enhanced Lung Function Testing: Adoption of oscillometry (forced oscillation technique) to measure respiratory system resistance and reactance, as a complementary tool of forced spirometry, exploring its potential for patients' monitoring and management of exacerbations.
2. Continuous Monitoring of IAQ at patients' homes: Assessment of advanced monitoring systems in patients' homes to continuously track air quality parameters, enabling the identification of environmental triggers linked to respiratory exacerbations.
3. Advanced Digital Support to innovative clinical processes with a two-fold aim: i) patient's empowerment for self-management of his/her condition, and ii) enhancing the role of the nurse case manager for early detection and management of exacerbations promoting share care agreements between the patient and the reference doctor (primary care physician and/or specialist). To this end, adoption of an Adaptive Case Management (ACM) Approach constitutes a key element.
4. Predictive Modeling: Development, and refinement, of machine learning-based modelling for early detection and management exacerbations. Key input data in the modelling approach will be: i) Clinical information (symptoms, Patient Reported Outcome Measures - PROMs), ii) Lung function testing, and iii) Patient's self-capturing physiological data through wrist sensors (health rate, heart rate variability and physical activity). Moreover, the impact of IAQ monitoring in the modelling will be explored.

The implementation, and refinement, of the four components alluded to above, as well as the design of the novel integrated care service, will be done with active engagement of patients, healthcare professionals, and other stakeholders in a co-design process using the Plan-Do-Study-Act (PDSA) methodology. Two PDSA cycles, with a six-month duration each, will be undertaken during 2024.

PHASE II (2025):

From January to December 2025, two additional PDSA cycles (six-month duration each) are planned to cover the following objectives:

1. Refinement of the novel integrated care service for enhanced management of exacerbations, as well as the implementation and continuous assessment of the four core components described in PHASE I.
2. Assessment of the outcomes of the novel integrated care service using the Quintuple Aim framework, that is, considering: i) Healthcare outcomes, ii) PROMs/Patient Reported Expirence Measures (PREMs), iii) healthcare professionals' engagement, iv) operational costs, and v) assessing equity. Comparison with conventional care will be done using a propensity score matching to elaborate a control group.
3. Evaluation of the process of deployment of the service using the Consolidated Framework for Implementation Research (CFIR) to identify barriers/facilitators for achieving a sustainable adoption, target candidates for the novel service, as well as potential for service transferability to other sites.

At the end of PHASE II, a mature service design ready for adoption should be available. Besides fulfilment of the objectives of K-Health in Air, the key lessons learned in the two-years period should provide novel insights for enhanced management of chronic patients with multimorbid conditions.

(Enclosed find: i) the Patient's Informed Consent approved by the Ethics Committee, as well as ii) the study protocol approved by the Ethics Committee of the Hosptial Clínic de Barcelona (HCB-2023-0126)).

ELIGIBILITY:
Inclusion Criteria:

* Aged Maximum 85 years
* Diagnosed with chronic obstructive pulmonary conditions such as COPD or treatment-resistant asthma.
* Exhibiting a high burden of co-morbidities, assessed above the 80th percentile of the regional risk stratification pyramid using Adjusted Morbidity Groups (AMG) scoring.
* Residing in Barcelona-Esquerra, except for treatment-resistant asthma patients, live in any district of the city of Barcelona.

Exclusion Criteria:

* Dementia.
* Inability to perform independent daily activities.

Max Age: 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study is recruiting 80% of participants from seven AISBE primary care facilities, each serving around 20,000 people. Recruitment leverages Catalan Health Surveillance System data to identify potential participants and link them with their primary care physicians, who engage with patients to assess participation willingness and ensure contact throughout follow-up. Initial contact involves a phone call from a nurse case manager to introduce the project and set up a home visit.
  The remaining 20% of the cohort, consisting of patients with treatment-resistant asthma, are recruited from the outpatient Severe Asthma Clinics at Hospital Clínic de Barcelona, using a similar approach.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-10-13 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Changes in use of healthcare resources - Unplanned hospital admissions | During 2025
  Number of unplanned hospital admissions.
  This outcome is part of a Quintuple Aim assessment of healthcare value generation of the novel integrated care service. Assessed in all individuals
Changes in use of healthcare resources - Exacerbations | During 2025
  Number and severity of exacerbations.
  This outcome is part of a Quintuple Aim assessment of healthcare value generation of the novel integrated care service. Assessed in all individuals
Changes in use of healthcare resources - Emergency room visits | During 2025
  Number of emergency room visits.
  This outcome is part of a Quintuple Aim assessment of healthcare value generation of the novel integrated care service. Assessed in all individuals
Changes in use of healthcare resources - Primary care visits. | During 2025
  Number of primary care visits.
  This outcome is part of a Quintuple Aim assessment of healthcare value generation of the novel integrated care service. Assessed in all individuals

SECONDARY OUTCOMES:
Healthcare costs | During 2025
  Healthcare costs in €
  This outcome is part of a Quintuple Aim assessment of healthcare value generation of the novel integrated care service. Assessed in all individuals
Patient reported experience (PREMs) - Enjoyment of life | During 2025
  Enjoyment of life: ICEpop CAPability measure for Older people (ICECAP-O)
  Scored on a scale from 0 to 1, where 0 represents no capability and 1 represents full capability.
  This outcome is part of a Quintuple Aim assessment of healthcare value generation of the novel integrated care service. It will be collected across the entire intervention group and in a randomly selected subset of 50 patients from the control group.
Patient reported experience (PREMs) - Resilience | During 2025
  Resilience: Brief Resilience Scale (BRS)
  Scores range from 1 to 5, with higher scores indicating greater resilience.
  This outcome is part of a Quintuple Aim assessment of healthcare value generation of the novel integrated care service. It will be collected across the entire intervention group and in a randomly selected subset of 50 patients from the control group.
Patient reported experience (PREMs) - Physical functioning | During 2025
  Physical functioning: 36-Item Short Form Survey (SF-36)
  Scores range from 0 to 100, where a higher score indicates better health status.
  This outcome is part of a Quintuple Aim assessment of healthcare value generation of the novel integrated care service. It will be collected across the entire intervention group and in a randomly selected subset of 50 patients from the control group.
Patient reported experience (PREMs) - Continuity of care | During 2025
  Continuity of care: Nijmegen Continuity Questionnaire (NCQ)
  Scores ranging on a Likert scale from 1 to 5.
  This outcome is part of a Quintuple Aim assessment of healthcare value generation of the novel integrated care service. It will be collected across the entire intervention group and in a randomly selected subset of 50 patients from the control group.
Patient reported experience (PREMs) - Physiological wellbeing | During 2025
  Physiological wellbeing: Mental Health Inventory-5 (MHI-5)
  Scored on a scale of 0 to 100, where higher scores indicate better mental health.
  This outcome is part of a Quintuple Aim assessment of healthcare value generation of the novel integrated care service. It will be collected across the entire intervention group and in a randomly selected subset of 50 patients from the control group.
Patient reported experience (PREMs) - Social Participation | During 2025
  Social Participation: Impact on Participation and Autonomy (IPA)
  Uses a scoring system based on a Likert scale ranging from 0 to 4 where higher scores indicate greater impairment in participation and autonomy.
  This outcome is part of a Quintuple Aim assessment of healthcare value generation of the novel integrated care service. It will be collected across the entire intervention group and in a randomly selected subset of 50 patients from the control group.
Patient reported experience (PREMs) - Person-centeredness | During 2025
  Person-centeredness: Patient Perceptions of Patient-Centeredness Questionnaire (P3CEQ)
  Typically uses a Likert scale from 1 to 5, with higher scores indicating better perceptions of patient-centeredness.
  This outcome is part of a Quintuple Aim assessment of healthcare value generation of the novel integrated care service. It will be collected across the entire intervention group and in a randomly selected subset of 50 patients from the control group.
Patient reported outcomes (PROMs) - Asthma symptoms | During 2025
  Asthma symptoms: Asthma Control Test (ACT)
  5 questions, each scored from 1 (poor control of asthma) to 5 (complete control of asthma). Higher scores indicate better asthma control.
  This outcome is part of a Quintuple Aim assessment of healthcare value generation of the novel integrated care service. It will be collected across the entire intervention group and in a randomly selected subset of 50 patients from the control group.
  *Depending on whether the primary disorder is asthma or COPD
Patient reported outcomes (PROMs) - Functional problems related to asthma | During 2025
  Functional problems related to asthma: Asthma Quality of Life Questionnaire (miniAQLQ)
  Designed to measure the functional problems (physical, emotional, social, and occupational) that are most troublesome to adults with asthma. It includes a series of questions scored from 1 (maximum impairment) to 7 (no impairment), with higher scores indicating better quality of life.
  This outcome is part of a Quintuple Aim assessment of healthcare value generation of the novel integrated care service. It will be collected across the entire intervention group and in a randomly selected subset of 50 patients from the control group.
  *Depending on whether the primary disorder is asthma or COPD
Patient reported outcomes (PROMs) - COPD symptoms | During 2025
  COPD symptoms: COPD Assessment Test (CAT)
  Each question is scored from 0 (no impact) to 5 (maximum impact), with the total score ranging from 0 (less impact) to 40 (more impact), indicating the severity of COPD.
  This outcome is part of a Quintuple Aim assessment of healthcare value generation of the novel integrated care service. It will be collected across the entire intervention group and in a randomly selected subset of 50 patients from the control group.
  *Depending on whether the primary disorder is asthma or COPD
Patient reported outcomes (PROMs) - Dyspnea | During 2025
  Dyspnea: Modified Medical Research Council (mMRC) Dyspnea Scale.
  It ranges from 0 (no breathlessness except with strenuous exercise) to 4 (too breathless to leave the house or breathless when dressing/undressing), with higher scores indicating more severe dyspnea.
  This outcome is part of a Quintuple Aim assessment of healthcare value generation of the novel integrated care service. It will be collected across the entire intervention group and in a randomly selected subset of 50 patients from the control group.
  *Depending on whether the primary disorder is asthma or COPD
Patient reported outcomes (PROMs) - Sino-Nasal symptoms | During 2025
  Sino-Nasal symptoms: Sino-Nasal Outcome Test (SNOT-22)
  22 items, each scored from 0 (no problem) to 5 (problem as bad as it can be). The total score can thus range from 0 (no sinus-related health problems) to 110 (severe sinus-related health problems).
  This outcome is part of a Quintuple Aim assessment of healthcare value generation of the novel integrated care service. It will be collected across the entire intervention group and in a randomly selected subset of 50 patients from the control group.
  *Depending on whether the primary disorder is asthma or COPD
Patient reported outcomes (PROMs) - Adherence to inhalers | During 2025
  Adherence to inhalers: Test of Adherence to Inhalers (TAI-12)
  12-item questionnaire used to assess a patient's adherence to inhaler medication in respiratory diseases. Each item is scored on a 5-point scale, with higher scores indicating better adherence. The total score ranges from 12 (poor adherence) to 60 (excellent adherence).
  This outcome is part of a Quintuple Aim assessment of healthcare value generation of the novel integrated care service. It will be collected across the entire intervention group and in a randomly selected subset of 50 patients from the control group.
  *Depending on whether the primary disorder is asthma or COPD
Equity of the intervention | During 2025
  Access to the service across different population groups: age, ethnicity, gender, socioeconomic status.
  This outcome is part of a Quintuple Aim assessment of healthcare value generation of the novel integrated care service. Assessed in all individuals
Performance of Predictive Modeling for Enhanced Management of Exacerbations | During 2025
  Model accuracy, sensitivity, specificity, positive predictive value, negative predictive value, and area under the receiver operating characteristic (ROC) curve
Performance of the digital support in terms of robustness and usability - Customer Satisfaction | During 2025
  Customer Satisfaction: Net Promoter Score (NPS)
  Measures customer loyalty and satisfaction. It is derived from asking customers a single question on a 0-10 scale
  Assessed in the intervention group only.
Performance of the digital support in terms of robustness and usability - Usability | During 2025
  Usability: System Usability Scale (SUS)
  Scored on a scale of 0 to 100, scores above 80 is an indicator of excellent usability, while a score below 60 could be problematic and suggests that the design needs improvements.
  Assessed in the intervention group only.

CONTACTS AND LOCATIONS:
Overall Officials: JOSEP ROCA TORRENT, MD, PHD, Principal Investigator — Institut d'Investigació Biomèdica August Pi I Sunyer (FRCB-IDIBAPS)
Locations (1):
- Fundació de Recerca Clínic Barcelona - Institut d'Investigació Biomèdica August Pi I Sunyer (FRCB-IDIBAPS), Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No
During the entirety of the project, it is not allowed to disseminate data. Nonetheless, should a formal request be submitted, it may be permissible to disclose certain elements of the information, albeit not in its totality.

REFERENCES:
- [Background] Herranz C, Martin-Moreno Banegas L, Dana Muzzio F, Siso-Almirall A, Roca J, Cano I. A Practice-Proven Adaptive Case Management Approach for Innovative Health Care Services (Health Circuit): Cluster Randomized Clinical Pilot and Descriptive Observational Study. J Med Internet Res. 2023 Jun 14;25:e47672. doi: 10.2196/47672. PMID 37314850
- [Background] Herranz C. A Co-Creation Process Toward Sustainable Adoption of Integrated Care for Prevention of Unplanned Hospitalizations. medRxiv. Published online January 1, 2023:2023.08.03.23293537. doi:10.1101/2023.08.03.23293537
- [Background] Veneroni C, Valach C, Wouters EFM, Gobbi A, Dellaca RL, Breyer MK, Hartl S, Sunanta O, Irvin CG, Schiffers C, Pompilio PP, Breyer-Kohansal R. Diagnostic Potential of Oscillometry: A Population-based Approach. Am J Respir Crit Care Med. 2024 Feb 15;209(4):444-453. doi: 10.1164/rccm.202306-0975OC. PMID 37972230
- [Background] Yamagami H, Tanaka A, Kishino Y, Mikuni H, Kawahara T, Ohta S, Yamamoto M, Suzuki S, Ohnishi T, Sagara H. Association between respiratory impedance measured by forced oscillation technique and exacerbations in patients with COPD. Int J Chron Obstruct Pulmon Dis. 2017 Dec 22;13:79-89. doi: 10.2147/COPD.S146669. eCollection 2018. PMID 29317813
- [Background] Wu CT, Li GH, Huang CT, Cheng YC, Chen CH, Chien JY, Kuo PH, Kuo LC, Lai F. Acute Exacerbation of a Chronic Obstructive Pulmonary Disease Prediction System Using Wearable Device Data, Machine Learning, and Deep Learning: Development and Cohort Study. JMIR Mhealth Uhealth. 2021 May 6;9(5):e22591. doi: 10.2196/22591. PMID 33955840
- [Background] Herranz C. An Adaptive Case Management Approach to Prevent Unplanned Hospital Admissions in a Care Continuum Scenario. Published online 2023.
- [Derived] Gomez-Lopez A, Arismendi E, Cano I, Farre R, Figols M, Hernandez C, Montilla-Ibarra A, Sanchez-Ruano N, Sanchez B, Siso-Almirall A, Sorribes M, Vela E, Piera-Jimenez J, Benavent J, Fermoso J, Roca J, Gonzalez-Colom R. Protocol for the enhanced management of multimorbid patients with COPD and severe asthma: role of indoor air quality. BMJ Open Respir Res. 2025 Jan 20;12(1):e002589. doi: 10.1136/bmjresp-2024-002589. PMID 39837595
- See also: EU PROJECT K-HEALTH IN AIR — https://k-healthinair.eu/
- See also: IDIBAPS Members of "Mecanismes fisiopatològics de les malalties respiratòries" — https://www.clinicbarcelona.org/ca/idibaps/arees-i-programes/biopatologia-i-bioenginyeria-respiratoria-cardiovascular-i-renal/mecanismes-fisiopatologics-de-les-malalties-respiratories/membres

DOCUMENTS (2):
  • Study Protocol (2023-11-30): https://cdn.clinicaltrials.gov/large-docs/02/NCT06421402/Prot_000.pdf
  • Informed Consent Form (2023-11-08): https://cdn.clinicaltrials.gov/large-docs/02/NCT06421402/ICF_001.pdf